CLINICAL TRIAL: NCT04624841
Title: Role of Indocyanine Green in Visualizing Critical View of Safety During Laparoscopic Cholecystectomy for Acute Cholecystitis
Brief Title: Indocyanine Green to Visualize Critical View of Safety During Laparoscopic Cholecystectomy for Acute Cholecystitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr Zia Ahmed Aftab, MBBS,FRCS,FACS, Consultant in Acute Care Surgery, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IRGC-05-NI-18-362; U1111-1256-1361 (Other: WHO International Clinical Trials Registry)
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Acute Cholecystitis; Acute; Cholecystitis, Choledocholithiasis; Acute Cholecystitis With Obstruction
Keywords: acute cholecystitis; laparoscopic cholecystectomy; critical view of safety; safe cholecystectomy; indocyanine green; operative cholangiogram; fluorescent imaging; near-infrared imaging
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis; Choledocholithiasis | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient is blinded to the intervention S/he receives. The surgeon, investigator, and outcomes assessor are masked but not strictly blinded up to the point when the near-infrared camera is switched on
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG group (Experimental): Participants receive an intravenous injection of 0.05 mg/kg of ICG 45 minutes preoperatively.
  A Pinpoint Endoscopic Fluorescence System (Novadac Technologies Inc., Canada) for ICG Fluorescence Observation with the easy switchable white light-fluorescent mode is used.
  Before dividing any tubular structure, the fluorescence imaging mode is routinely used again, and fluorescent angiography is performed by re-injecting the same dose of ICG as initially used.
  After the division of the cystic duct and artery, the fluorescence imaging mode is applied again to check for bile leakage.
  Interventions: Drug: Indocyanine Green
- No ICG Group (No Intervention): No ICG is administered after randomization of the patient to a control group and hence will not produce any enhancement of the image on A Pinpoint Endoscopic Fluorescence System for ICG Fluorescence Observation. This will continue as a routine Laparoscopic cholecystectomy without fluorescent imaging enhancement.

INTERVENTIONS:
Drug: Indocyanine Green — 2.5-7.5 mg (0.05 mg/kg) injection
  Other Names: ICG; fluorescent Imaging
  Arms: ICG group

SUMMARY:
The purpose of this prospective randomized trial is to study the role of Indocyanine green (ICG) to visualize the Critical View of Safety during emergency Laparoscopic Cholecystectomy for patients with Acute Cholecystitis.

DETAILED DESCRIPTION:
After informing about the study and obtaining consent to participate, patients who are diagnosed with Acute Cholecystitis and posted for emergency Laparoscopic Cholecystectomy will be randomly assigned to receive either ICG or not as a method to identify the Critical View of Safety during the operation.

The primary outcome is whether there was a precise and satisfactory visualization of the junction between the cystic duct, the common hepatic duct, and the common bile duct by indocyanine green compared to the control group. The time taken to achieve this will be measured in minutes from video recordings of the laparoscopic surgery. The process will be further assessed by a surgeons' satisfaction score.

The expected duration of the study will be 12 months involving a total of 80 patients randomized into two groups- 40 patients in the intervention group and 40 patients in the control group.

The expected outcome of the study is that ICG is more effective than the control group in providing precise and satisfactory visualization of Critical View of Safety and takes less time. We predict the surgeons to be equally or more satisfied with ICG compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for emergency Laparoscopic Cholecystectomy for Acute Cholecystitis
* Patient age ≥ 18 years.
* Patients who consent to take part in the study

Exclusion Criteria:

* Preoperative planned for Open Cholecystectomy
* Allergy towards iodine, iohexol or ICG
* Pregnancy or lactation
* Renal insufficiency
* Legally incompetent for any reason
* Withdrawal of inclusion consent at any time
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of surgeries in which Critical View of Safety was achieved | Prior to clipping of the Cystic Duct and Cystic Artery or decision to perform conventional intraoperative cholangiography or convert to open.
  Percentage of surgeries where there was complete visualization of Critical View of Safety by intraoperative fluorescent cholangiography compared to the control group with no fluorescent imaging. Complete visualization of the Critical View of Safety is defined by the SAGS guidelines.
  The laparoscopic procedure is recorded & assessed individually & separately by two consultant surgeons who are not the operating surgeon whether the Critical View of Safety was achieved prior to clipping of Cystic Duct & Cystic Artery.
  Failure of identification of Critical View of Safety is defined as the need for further conventional intraoperative cholangiography or open conversion due to inability to accurately identify the biliary anatomy to complete the cholecystectomy safely.

SECONDARY OUTCOMES:
Time taken to identify Critical View of Safety | After securing working ports till Clipping of Cystic Duct or Artery.
  Time taken by intraoperative fluorescent cholangiography or control group to identify Critical View of Safety. The laparoscopic procedure is recorded and Time taken is recorded by the Primary Investigator as the total time between successful introduction of the operative ports until the Critical View of Safety is achieved and Cystic Duct and Cystic Artery are clipped.
Surgeon's Satisfaction Survey | Prior to clipping of the Cystic Duct and Cystic Artery or decision to perform conventional intraoperative cholangiography or convert to open.
  Surgeon satisfaction survey will be completed by the operating surgeon intraoperatively by answering the question "Are you satisfied to proceed with the laparoscopic cholecystectomy without a conventional intraoperative cholangiography?". The answers will be a binary Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Zia Aftab, MBBS, FACS, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishizawa T, Bandai Y, Kokudo N. Fluorescent cholangiography using indocyanine green for laparoscopic cholecystectomy: an initial experience. Arch Surg. 2009 Apr;144(4):381-2. doi: 10.1001/archsurg.2009.9. No abstract available. PMID 19380655
- [Background] Daskalaki D, Fernandes E, Wang X, Bianco FM, Elli EF, Ayloo S, Masrur M, Milone L, Giulianotti PC. Indocyanine green (ICG) fluorescent cholangiography during robotic cholecystectomy: results of 184 consecutive cases in a single institution. Surg Innov. 2014 Dec;21(6):615-21. doi: 10.1177/1553350614524839. Epub 2014 Mar 9. PMID 24616013
- [Background] Dip F, Roy M, Lo Menzo E, Simpfendorfer C, Szomstein S, Rosenthal RJ. Routine use of fluorescent incisionless cholangiography as a new imaging modality during laparoscopic cholecystectomy. Surg Endosc. 2015 Jun;29(6):1621-6. doi: 10.1007/s00464-014-3853-7. Epub 2014 Oct 3. PMID 25277476
- [Background] Pesce A, Piccolo G, La Greca G, Puleo S. Utility of fluorescent cholangiography during laparoscopic cholecystectomy: A systematic review. World J Gastroenterol. 2015 Jul 7;21(25):7877-83. doi: 10.3748/wjg.v21.i25.7877. PMID 26167088
- [Background] Overby DW, Apelgren KN, Richardson W, Fanelli R; Society of American Gastrointestinal and Endoscopic Surgeons. SAGES guidelines for the clinical application of laparoscopic biliary tract surgery. Surg Endosc. 2010 Oct;24(10):2368-86. doi: 10.1007/s00464-010-1268-7. Epub 2010 Aug 13. No abstract available. PMID 20706739